CLINICAL TRIAL: NCT05226988
Title: The Study Firstly Proposes a Hybrid Robot-assisted Training Program, Which Combines Two Types of Robotic Systems, to Enhance the Effectiveness of Robot-assisted Training and Provide a New Approach for Motor Training of Upper Limb in Stroke Patients
Brief Title: Effect of Hybrid Robot-assisted Training Using End-effector and Exoskeleton Devices in Distal Upper Extremity After Stroke：Motor Control, Motor and Daily Function, Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202101742B0
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: neurorehabilitation; robot-assisted training; upper extremity; motor control
MeSH Terms: conditions — Stroke | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hybrid-RT (Experimental): hybrid robot-assisted training
  Interventions: Device: robot-assisted
- Exo-RT (Experimental): exoskeleton robot-assisted training
  Interventions: Device: robot-assisted
- EE-RT (Experimental): end-effector robot-assisted training
  Interventions: Device: robot-assisted
- conventional training groups (Active Comparator)
  Interventions: Device: Conventional rehabilitation intervention

INTERVENTIONS:
Device: robot-assisted — Participants received the 18-session robot-assisted intervention 3 sessions a week for 6 consecutive weeks. Each session consisted of 20-minute continuous passive motion, 20-minute active motion practice, and 30-minute task-oriented practice.
  Arms: EE-RT; Exo-RT; Hybrid-RT
Device: Conventional rehabilitation intervention — Participants received the 18-session conventional rehabilitation intervention 3 sessions a week for 6 consecutive weeks. The intervention consisted of warm up including range of motion exercise, and strengthening exercise followed by task-oriented training for activities of daily living.
  Arms: conventional training groups

SUMMARY:
The purpose of this study is to examine the immediate and long-term effects of hybrid robot-assisted training (Hybrid-RT), exoskeleton robot-assisted training (Exo-RT), end-effector robot-assisted training (EE-RT), and conventional training on stroke patients' motor performance, daily life functions, quality of life, and self-efficacy.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability, and most stroke survivors have chronic upper limb dysfunction, which affects participation in activities of daily living. In addition to conventional rehabilitation training, robot-assisted training has been advocated as a contemporary approach of hand function training. Robotic devices can be categorized into exoskeleton and end-effector types based on their mechanical design. However, previous studies did not reach an agreement on the effectiveness of two types of robot-assisted training. The study firstly proposes a hybrid robot-assisted training program, which combines two types of robotic systems, to enhance the effectiveness of robot-assisted training and provide a new approach for motor training of upper limb in stroke patients. Secondly, the relative effects of the two types of robot-assisted training will be compared. The purpose of this study is to examine the immediate and long-term effects of hybrid robot-assisted training , exoskeleton robot-assisted training , end-effector robot-assisted training , and conventional training on stroke patients' motor performance, daily life functions, quality of life, and self-efficacy. The study will recruit stroke patients and randomly assign them to the hybrid robot-assisted training, exoskeleton robot-assisted training, end-effector robot-assisted training, and conventional training groups. Each participant will receive training 3 sessions a week for 6 consecutive weeks. Participants will be assessed at baseline, after the intervention, and at 3-month follow-up. Repeated measures of analysis of variance will be used to evaluate the changes within each intervention group at three evaluation times and to compare the differences between the four intervention groups. In order to understand the motor learning effects after receiving different interventions, the investigator use kinematic analysis to investigate the movement control mechanism of upper limb movements. The findings of this study will build the evidence-based foundation for bridging the gap between basic science and clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Stroke more than 3 months.
* Modified Ashworth Scale proximal part ≤ 3, Modified Ashworth Scale distal part ≤ 2, and no serious muscle spasms.
* The myoelectric signal can be detected to activate the instrument
* Unilateral paresis (FMA score<60)
* No serious cognitive impairment (i.e., Mini Mental State Exam score > 24)
* Can provide informed consent

Exclusion Criteria:

* Other neurological disease
* Complete sense of body defect
* Inability to understand instructions
* current participation in any other research
* Botulinum Toxin injection within 3 months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Change scores of Fugl-Myer Assessment (FMA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The upper-extremity subscale of the FMA will be used to assess motor impairment. There are 33 upper extremity items measuring the movements and reflexes of the shoulder/elbow/forearm, wrist, hand, and coordination/speed. Each score is on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully). The maximum score is 66, indicating optimal recovery. The subscore of a proximal shoulder/elbow (FMA s/e: 0-42) and a distal hand/wrist (FMA h/w: 0-24) will be calculated to investigate the treatment effects on separate upper extremity elements. The FMA has good reliability, validity, and responsiveness in stroke patients.
Change scores of Active Range of Motion (AROM) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Patient performs the exercise to move the joint without any assistance to the muscles surrounding the joint.
Change scores of grip and pinch power | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Jamar hand dynamometer is the most widely cited in the literature and accepted as the gold standard by which other dynamometers are evaluated. Excellent concurrent validity of the Jamar hand dynamometer is reported. The Jamar hand dynamometer measure the grip-strength. The norm of healthy male aged 18 to 75 years is from 64.8 lb to 121.8 lb, while the norm of healthy female aged 18 to 75 years is from 41.5 lb to 78.7 lb. Higher value represent a greater grip-strength.
Change scores of Modified Ashworth (MAS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Modified Ashworth Scale is a 6-point (0、1、1.5、2、3、4) ordinal scale that measures muscle spasticity in patients with brain lesions. Higher score indicates higher muscle tone. Investigators will assess the Modified Ashworth Scale scores of UE muscles, including biceps, triceps, wrist flexors and extensors, and finger flexors and extensors. The validity and reliability of Modified Ashworth Scale for patients with stroke were established to be adequate to good.
  The total score of Modified Ashworth ranged from 0 to 32.
Change scores of Medical Research Council (MRC) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Medical Research Council is an ordinal scale that assesses muscle strength. The scoring for each muscle ranges from 0 to 5, with a higher score indicates stronger muscle. The reliability of Medical Research Council for all muscle groups was good to excellent in patients with stroke.
  The total score of Medical Research Council ranged from 0 to 20.
Change scores of Revised Nottingham Sensory Assessment (rNSA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The rNSA includes tactile sensation, kinesthetic sensation, and stereognosis. The rNSA is reliable measure of sensory function in stroke patients. For tactile sensation, the patient will be asked to indicate whenever he or she feels the test sensation. For kinesthetic sensations, all 3 aspects of movement will be tested: appreciation of movement, its direction and accurate joint position sense. The limb on the affected side of the body will be supported and moved by the examiner in various directions but movement is only at one joint at a time. The patients will be asked to mirror the change of movement with the other limb. For stereognosis, the object will be placed in the patient's hand for a maximum of 30 seconds. Identification is by naming, description or by pair-matching with an identical set. The object may be moved around the affected hand by the examiner. The rNSA has good intrarater and interrater reliability.
Change scores of Wolf Motor Function Test (WMFT) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The WMFT was designed to assess the effects of CIT on arm function after stroke and traumatic brain injury (Wolf, Lecraw, Barton, & Jann, 1989). There are 15 function-based and 2 strength-based tasks. For timed functional tasks, completion times from 0 to 120 seconds are averaged. For functional ability scoring, 6-point ordinal scales are used, where 0 indicates "does not attempt with the involved arm" and 5 indicates "arm does participate, movement appears to be normal." The clinimetrics of the WMFT has been ascertained in stroke patients.
Change scores of Mini-Mental State Exam (MMSE) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of Montreal Cognitive Assessment (MoCA) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitvie functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Motor Activity Log (MAL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The MAL consists of 30 structured questions to interview how the patients rate the frequency (amount of use subscale) and quality (quality of movement subscale) of movements while using their affected arm to accomplish each of the 30 daily activities. The score of each item ranges from 0 to 5, and the higher scores indicate more frequently used or higher quality of movements. The clinimetric properties of the MAL in stroke patients have been validated
Change scores of Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The NEADL scale is a measure of Instrumental ADL ability, comprising sub-scales for mobility, household ability and leisure activity. The NEADL consists of 22 activity items, scoring on the basis of the required level of assistance. The range of total score is 0-66, and higher score representing better function. This measure is administered 3 times during the study period.
Change scores of Stroke Impact Scale (SIS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. The reliability, validity, and responsiveness have been shown to be satisfactory in stroke patients.
Change scores of stroke self-efficacy questionnaire (SSEQ) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  the Stroke Self-Efficacy Questionnaire (SSEQ) , a questionnaire developed to measure the most relevant self-efficacy and self-management domains specific to the stroke population. It contains 13 items that are rated on a 0 - 10 scale, with higher scores indicating greater levels of self-efficacy. Questionnaire includes a range of relevant functional tasks such as walking, getting comfortable in bed, as well as some self-management tasks.
Change scores of Daily Living Self-Efficacy Scale (DLSES) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The DLSES is designed to measure self-efficacy in psychosocial functioning and self-efficacy in activities of daily living, regardless of level of physical impairment.
Change scores of Functional Abilities Confidence Scale (FACS) | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The Functional Abilities Confidence Scale (FACS) was designed to measure the degree of self-efficacy or confidence a patient exhibits with various movements or postures.
Kinematic analysis | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.
Change scores of pain threshold measurements | Baseline, post test immediately after completing 18 intervention sessions (around 6 weeks after baseline), follow up test (3 months after completing intervention sessions)
  Devices that apply and simultaneously measure pressure to evoke pain are called 'pressure algometers,' which are usually pistol-shaped with an operator handle and a single protruding probe that is applied to the subject's body surface.
  Pressure stimuli are ordinarily applied at static, individual sites when using algometers. Nevertheless, other loading regimens are feasible: moving the site of pressure while loaded, using a wheel probe or a sliding probe ; multiple site stimulation through gripping opposite sides of a digit , or an inflatable tourniquet cuff that applies circumferential pressure around an entire limb .

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan